CLINICAL TRIAL: NCT04235556
Title: Integrated Management of Care Pathway in Oncology. Impact on the Delay of Therapeutic Management and the Satisfaction of Patients and Carers
Brief Title: Integrated Care Pathway in Oncology (PASSION)
Acronym: PASSION
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: MSD France (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP190973
Record Dates: First submitted 2019-12-02; First posted 2020-01-22 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer; Gastric Cancer; Pancreatic Cancer; Thoracic Neoplasms; Breast Cancer; Ovarian Cancer; Bladder Cancer; Prostate Cancer
Keywords: care pathway; satisfaction; oncology; treatment delay
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Thoracic Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Personal Satisfaction; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historic cohort: Retrospective cohort of patients that were treated in the Hôpital Européen Georges Pompidou before the creation of the care pathway unit.
- Prospective cohort: All consecutive patients that meet the inclusion criterion and will begin a cancer care after the study start.
  Interventions: Behavioral: Care pathway unit

INTERVENTIONS:
Behavioral: Care pathway unit — Patients from the prospective cohort will have their health care scheduled by the care pathway unit.
  Groups: Prospective cohort

SUMMARY:
A centralized unit for integrated management of care pathway in Oncology has been created. This unit settles the patients' appointments (biopsy, intravenous device, chemotherapy, imaging, oncologist...).

The aim of this study is to assess the delay between the first appointment with the oncologist and the beginning of the antitumoral treatment, and therefore evaluate the efficacy of the care pathway unit.

The second aim is to assess the satisfaction of patients and health care teams.

DETAILED DESCRIPTION:
PASSION is a french monocentric study.

For the retrospective cohort, patient will be selected through the use of data warehouse available on the HEGP.

For the prospective cohort, patient will be included according to the selection criteria.

Each patient will be followed up during 6 month and a satisfaction questionnaire will be completed at 1 month and 4 month of the first administration of anti-tumor therapy.

For both cohort, clinical-anatomo-biological data will be collected through the use of data warehouse available on the HEGP.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven : colon, gastric, pancreatic, prostate, bladder, breast, thoracic, or ovarian cancer
* First appointment for cancer care at the Hôpital Européen Georges Pompidou
* Intravenous antitumoral treatment

Exclusion Criteria:

* Medical care non covered by social welfare
* Radiochemotherapy
* Death in the 6 months following first oncological appointment or absence of medical care in the year following the first oncological appointment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort: patients treated at the Hôpital Européen Georges Pompidou in 2015 and 2017.
  Prospective cohort:
  * Histologically proven : colon, gastric, pancreatic, prostate, bladder, breast, thoracic, or ovarian cancer
  * First appointment for cancer care at the Hôpital Européen Georges Pompidou
  * Ile de France resident
  * All appointments planned at the Hôpital Européen Georges Pompidou
  * Intravenous antitumoral treatment
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time between the first appointment with the oncologist and the beginning of antitumoral treatment. | 6 months
  Delay of health care

SECONDARY OUTCOMES:
Patients satisfaction | 6 months
  Satisfaction of patients with OUT-PATSAT35 questionnaire (out-patient satisfaction) : Likert type scale with 5 ordered modalities (bad to excellent), rated from 1 to 5.
Health care teams satisfaction | 6 months
  Satisfaction of health care teams : qualitative questionnaire with 4 ordered modalities (very satisfied to not satisfied)
Rate of emergency consultations and hospitalizations | 6 months
  Need for unexpected health care

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Bichon, Principal Investigator — AP-HP, Hôpital Européen Georges Pompidou, Paris
Locations (1):
- AP-HP Hôpital européen Georges-Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: one year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization